CLINICAL TRIAL: NCT00594009
Title: Safety and Efficacy of Venovenous Carbon Dioxide Removal in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Acute Respiratory Failure (ARF)
Brief Title: Venovenous CO2 Removal (VVCO2R) in Patients With COPD and Acute Respiratory Failure
Acronym: VVCO2R
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to loss of key personnel due to illness and sabbatical of thePI
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-142
Record Dates: First submitted 2007-12-17; First posted 2008-01-15 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2015-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venovenous CO2 Removal (VVCO2R) in COPD (Experimental): All patients enrolled in the trial will receive VVCO2R which consists of a circuit with a centrifugal pump, tubing, double lumen intravenous catheter and hollow fiber oxygenator
  Interventions: Device: Venovenous CO2 Removal (VVCO2R) in COPD

INTERVENTIONS:
Device: Venovenous CO2 Removal (VVCO2R) in COPD — Patients who meet criteria will be placed on an extracorporeal circuit consisting of an oxygenator, centrifugal pump, tubing and indwelling double lumen venous catheter for CO2 removal for up to 96 hours for treatment of COPD exacerbation requiring hospitalization and intensive care
  Other Names: (VVCO2R)

SUMMARY:
The purpose of this study to determine the safety and effectiveness of a mechanical device to remove carbon dioxide from the blood of patients with chronic obstructive pulmonary disease (COPD)when they are hospitalized in the intensive care unit for exacerbation of their condition.

DETAILED DESCRIPTION:
This is a pilot study to examine the efficacy and safety of an extracorporeal circuit to remove carbon dioxide (CO2) from the blood in patients with an acute exacerbation of COPD resulting in acute or acute on chronic respiratory failure. The extracorporeal circuit consists of venovenous configuration through a percutaneously inserted 18 F double lumen catheter placed in a central vein. Centrifugal pump and heparin bonded circuit are used and patient is heparinized to maintain an activated clotting time (ACT) > 180. Circuit blood flow and gas sweep speed will be adjusted to maximize CO2 removal and minimize ventilator settings and patient's work of breathing. Patients will remain on the extracorporeal circuit for a maximum of four days as tolerated. Plasma Hemoglobin will be monitored daily.

ELIGIBILITY:
Inclusion Criteria:

1. Acute respiratory failure on invasive mechanical ventilation or
2. Acute respiratory failure and an advanced directive foregoing invasive mechanical ventilation
3. Established diagnosis of COPD
4. Age group: 18 years or greater

Exclusion Criteria:

1. Significant vasopressor support
2. Systolic BP < 100 torr systolic despite vasopressor support
3. Class III or Class IV congestive heart failure
4. Left ventricular ejection fraction < 30% by previous echocardiogram
5. Recent (6 month) history of myocardial infarction
6. Coronary artery disease with unstable angina
7. Recent (6 month) history of venous embolism
8. Uncontrolled coagulopathy (international normalized ratio (INR) > 5 or activated partial thromboplastin time (aPTT) > 80s) despite corrective therapy
9. History of heparin-induced thrombocytopenia or other adverse event following the administration of heparin (heparin group only)
10. Pregnancy
11. Severe chronic liver disease
12. Severe anemia (Hgb < 9 gm/dl)
13. Any contraindication to systemic anticoagulation with heparin, including recent central nervous system injury or hemorrhage, retinal hemorrhage or other recent hemorrhage from sites which cannot be controlled
14. Technically unable to access vessels (obesity, limb deformity, previous surgery at the site, infection, etc.)
15. Evidence of increased intracranial pressure or history of an intracranial hemorrhage within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor J Cardenas, Jr, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Venovenous CO2 Removal (VVCO2R) in COPD: All patients enrolled in the trial will receive the proposed Patients who meet criteria will be placed on an extracorporeal device for CO2 removal for up to 96 hours for treatment of COPD exacerbation requiring hospitalization and intensive care
Period: Overall Study
Arm/Group | Venovenous CO2 Removal (VVCO2R) in COPD
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- VVCO2R in COPD: All patients enrolled in the trial will receive the proposed intervention
  Rotaflow centrifugal pump (Maquet, Inc.): Patients who meet criteria will be placed on an extracorporeal device for CO2 removal for up to 96 hours for treatment of COPD exacerbation requiring hospitalization and intensive care
Arm/Group | VVCO2R in COPD
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (NA) — only one subject
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
chronic obstructive pulmonary disease (COPD) patients [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: The Amount of CO2 Transferred Through the Oxygenator at Various Levels of Blood and Gas Flow
Description: The amount of CO2 removed in cc/min will be recorded. The level of blood flow (ml/min) and gas flow (l/min) at each measurement of CO2 removal will also be recorded
Time Frame: 0 to 96 hours
Measure: Number; unit: cc/min
Groups:
- VVCO2R in COPD: All patients enrolled in the trial will receive the proposed intervention
  Patients who meet criteria will be placed on an extracorporeal device for CO2 removal for up to 96 hours for treatment of COPD exacerbation requiring hospitalization and intensive care
Arm/Group | VVCO2R in COPD
Number analyzed (Participants) | 1
cc/min | 75

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study period and up to 14 days after discontinuation of device
Arm/Group | VVCO2R in COPD
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes